CLINICAL TRIAL: NCT05655026
Title: The Use of Non-invasive Respiratory Assistance to Facilitate Bronchofiberoscopy Performance in Patients With Hypoxemic (Type One) Respiratory Failure
Brief Title: NIV-FOB, HFNC-FOB- Comparison of Methods
Acronym: NIRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2202
Record Dates: First submitted 2022-06-15; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-06

CONDITIONS: Respiratory Failure; Hypoxemia; Hypoxemic Respiratory Failure
Keywords: respiratory failure; non invasive ventilation; bronchofiberoscopy
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- x≤300 HFNO or standard oxygen supplementation (Experimental): bronchoscopy, taking blood gas, taking blood for blood test
  Interventions: Device: NIV, HFNO
- 100<x≤200 NIV or HFNO (Experimental): bronchoscopy, taking blood gas, taking blood for blood test
  Interventions: Device: NIV, HFNO
- x≤100 NIV or intubation (Experimental): bronchoscopy, taking blood gas, taking blood for blood test, intubation
  Interventions: Device: NIV, HFNO

INTERVENTIONS:
Device: NIV, HFNO — Arterial blood pressure and saturation will be measured. Arterial blood gases will be collected to qualify patients to one of the three groups. After qualification, patient will be randomly assigned to a given respiratory support method during FB.

SUMMARY:
The aim of the study is to asses safety and indications and contraindications for performing bronchofiberocopy (FB) with respiratory support methods, i.e. non-invasive ventilation (NIV) and high flow nasal oxygen therapy (HFNO). Additionally, researchers want to determine how using these methods could avoid the risk of most common complications such as: hypoxemia-related events, decompensation of chronic respiratory failure, worsening of gas exchange, hemodynamic instability.

DETAILED DESCRIPTION:
Bronchofiberoscopy (FOB) is a minimally invasive procedure that has been commonly performed for many years in pneumological patients and in patients requiring intensive medical care.inistered to let patients tolerate FOB is an additional factor for derangement of blood gases. FB is usually performed with oxygen supplementation administered through standard nasal cannula. Due to increasing number of seriously ill, patient with respiratory failure, pure oxygen support is frequently insufficient to assure accurate oxygenation and prevent hypercapnia in patients requiring FOB. Up till now, many of those patients have been disqualified or intubated from FOB due to unfavorable risk to benefits balance.

NIV assures normal minute ventilation in patients with decreased respiratory drive, prevents collapsing of the peripheral airways, prevents atelectasis development, facilitates alveoli recruitment, increases vital capacity and lung susceptibility, as well as decrease heart workload. NIV may enable therapeutic FOB performance in patients with alveolar proteinosis without the need for intubation. NIV allows to perform safe bronchofiberoscopy in both diagnostic and therapeutic indications in patients with exacerbation of respiratory failure as well as in patients with severe chronic respiratory failure.

HFNC is another innovative method of respiratory support, which generates turbulent flow in patient's nasopharyngeal cavity and facilitates precise settings of high oxygen concentrations FiO2 up to 1 (100%). Obtained high flow is associated with generation of positive airway pressure, which additionally recruits alveoli and reduces atelectasis, which is partially similar to NIV and may give additional benefits to treatment of respiratory failure. Preliminary data indicate that both of described methods have a potential role in increasing the safety of FOB examinations in patients with mild to moderate respiratory failure. However, as of today it has not been clearly supported by scientific evidence, whether there are differences in the indications, contraindications, complications risk. As so far there is lack of evidence which would clearly indicate the target population which would benefit mostly from NIV-FOB or HFNC-FOB.

Additionally, investigators do not currently know universal settings of both devices which could be used initially and universally during FOB in patients with different severity of respiratory failure. In patients with severe respiratory failure, in some cases it is compulsory to intubate patient in order to perform a safe bronchoscopy. In cases of patient who have not been intubated, FOB could cause exacerbation of underlying respiratory failure, which may require intubation and ICU transfer.

This is a multicenter international three-arm Randomized Controlled Trial (RCT) performed in departments which deal with patients suffering from respiratory failure: respiratory intensive care unit (RICU), bronchoscopic theatre- form patients treated in other departments such as internal medicine departments, cardiology etc, pulmonary ward and ICU departments in apriori not intubated patients.

Patient will be assigned to each study arm based on Horowitz index calculated on the basis of the pO2 results obtained from arterial blood gas test and FiO2 during the study. In each arm, patient will be randomly assigned to one from dwo dedicated respiratory support methods.

To assess the best and safe indication for performing FOB with different levels of respiratory support according to escalating degrees of severity of blood gases derangements.

The topic of study is clinically important because defining precise indications for the use of NIV or HFNC during FOB, could facilitate FOB performance in a larger group of patients, which would initially be disqualified from this procedure. Additionally, it probably may reduce the group of patients who would require intubation for FOB performance. Moreover, the use of HFNC or NIV may probably decrease the FOB and sedation related risk.

The aim of study:

* Verification of the role of HFNC and NIV in increasing FOB safety gained by preventing FB correlated complications,
* Determination of indications for non-invasive respiratory assistance (HFNC-FOB, NIV-FOB) facilitated -FOB and FOB under mechanically invasively ventilated patient (MV-FB) according to criteria of escalating in the severity of type one respiratory failure under FB,
* Determination of optimal settings of HFNC and NIV during FOB,
* Taking into account oxygenation criterion used to identify ARDS severity we have decided to use the Berlin ARDS criteria cut-off points to choose to perform FB under either O2 vs HFNC, HFNC VS NIV or NIV VS IMV. CPAP - was not included into the study arms, because although it improves oxygenation is generally not accepted as a ventilation mode, because it does not generate pressure support but eventual increased work of breathing is caused by reduced work of breathing and alveolar recrutation. Moreover, HFNC has the potential to generate PEEP on a level of about 5 cmH2O. Lastly most machines used nowadays in bronchoscopy labs have both NIV and CPAP mode therefore it seems more accurate to use the NIV settings which theoretically should be more effective and safer in sedated patients.

The target number of 300 patients in all groups (100 patients in each) was calculated on the basis of intubation risk in patients with respiratory failure which is reported to be on the level between 0.2-2%.

Methodology Before FB A detailed medical history (including comorbidities, pharmacotherapy, smoking history and NYHA, mMRC, Charlson, BORG, Apache II, SAPS II, RASS-will be assessed during FB scales) will be collected. Lung function test (spirometry) and 6-minutes walking test (6MWT) will be performed if only possible due to patients' clinical condition. Arterial blood pressure and saturation will be measured. Arterial blood gases will be collected to qualify patients to one of the three groups. After qualification, patient will be randomly assigned to a given respiratory support method during FB.

Procedure and rescue escalated support HFNC or passive oxygen therapies will be used with dedicated nasal cannulas. NIV will be performed with a dedicated bronchoscopic interface with bronchoscopic elbow. The study will compare the initial settings of the devices, which will be maintained if possible based on clinical condition of the patient. In the case of desaturation, hypercapnia or other abnormalities in the patient's clinical condition, the device settings may be changed according to the protocol or the method may be upgraded (HFNC->NIV->MV).

Monitoring During FOB: FiO2, TcCO2, ECG and heart rate (constant assessment) and arterial blood pressure (every 5 minutes) will be assessed.

After FOB After FOB arterial blood gases will be collected again and possible complications will be reported (bronchospasm, hypoxemia, decompensated respiratory acidosis, local bleeding, fever, premature termination of examination, ICU transfer, pneumothorax, death). FOB will be performed with a use of: optic,video or EBUS bronchofiberoscopes. The outer diameter of used bronchoscope should be reported. The type and dosage of sedatives should be reported in all study arms; however, dedication sedation depth should target RASS -2 to -3.

The data obtained from the interview and additional results will be entered anonymously and in compliance with GDPR criteria into computer database and statistically processed.

Support device settings

1. Standard oxygen: 3L/min increased up till 10L/min to maintain SaO2>92%,
2. HFNC: flow 60L/min, temp 34C, and oxygen supplementation (FiO2) adjusted to maintain SaO2≥ 92%,
3. NIV will be conducted in the spontaneous timed (ST) mode, with a backup rate of 16-18 per min, Tins 0,8-1s, expiratory positive airway pressure (EPAP) of 6-16 cmH2O, pressure support (PS) of 8-30 cmH2O and the oxygen supplementation titrated to maintain SaO2≥ 92%,
4. IMV: The ventilator settings initially will match the previous settings to keep the SaO2≥ 92, based on minute ventilation and tidal volume. The detailed initial mode, as well as settings including PS and EPAP, FiO2 should be reported. In intubated patients: intubation tube size, should be recorded,
5. In cases of all devices the patient will have 5-15 minutes for acclimatization before the bronchoscopy starts.

The primary general expected endpoints

* Possibility to perform (therapeutic and/or diagnostic) FB in patients who would otherwise be disqualified or intubated,
* Improvement of patient's comfort during the examination (possibility to use deeper sedation)
* Increased safety and comfort of FB in patients with respiratory failure (decreased number of procedure related both benign and severe complications).

The primary specific assessed endpoints:

1. Hypoxemia >5% SaO2 fall, longer than 30 seconds,
2. Hypercapnia >5mmHg CO2 increase longer than 30 seonds,
3. New onset of cardiac arrythmia,
4. Hypotension below 90/60 or more than 30% of initial level,
5. The need for escalation of treatment O2-to HFNO to NIV-to intubation,
6. Transfer to ICU,
7. Resuscitation,
8. Intubation,
9. Death.

All complications described in 3 categories (1- directly during bronchoscopy, within 2 hours from the termination of bronchoscopy and happening within 24 hours from the procedure)

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years, with indications for bronchoscopy,

   * Diagnostic procedure: lung cancer, hemoptysis, BAL in interstitial lung diseases.
   * Therapeutic procedure: pneumonia in patients with impaired cough reflex, performed to obtain sputum cultures and bronchial tree toilet, hemoptysis or foreign body aspiration in patients not requiring rigid bronchoscopic management.
2. Written informed consent to participate in the study,
3. PO2/fiO2≤300 in blood gas test performed directly (within 24 h) during the qualification for FB

Exclusion Criteria:

1. No willingness to participate,
2. PO2/fiO2>300 in arterial blood gases, severe unstable coronary artery disease (CCS III/IV), NYHA III/IV,
3. Hemodynamic instability defined as continuous amine influx. Myocardial infarction during the last 2 weeks, without PCI treatment. Unstable angina, severe arrhythmias - especially ventricular,
4. Chronic primary pulmonary hypertension confirmed by right heart catherisation in WHO III/IV,
5. Unsecured by chest tube pneumothorax,
6. Platelet count <20,000 /µl (without platelet transfusion),
7. INR >2 or APTT >36 s., in case of diagnostic FB [18]
8. The study will also not include patients who were intubated before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Hypoxemia | 2 years
  measure by pulsoxymetry, blood gas test. Number of Participants with procedure related complications
Comfort | 2 years
  Use dedicated questionaire to asses patient condition after bronchoskopy
Safety | 2 years
  Number of Participants with procedure related complications

CONTACTS AND LOCATIONS:
Locations (1):
- Aleksandra, Katowice, Poland

IPD SHARING:
Plan to Share IPD: No
Including other hospitals. Speech at the conference. Prepare manuscript.